CLINICAL TRIAL: NCT02021825
Title: Efficacy and Safety of Mitoxantrone in Patients With Refractory Neuromyelitis Optica and Spectrum Disorders
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MITONMO
Record Dates: First submitted 2013-09-03; First posted 2013-12-27 (Estimated); Last update posted 2013-12-27 (Estimated); Status verified 2013-12

CONDITIONS: Neuromyelitis Optica; Neuromyelitis Optica Spectrum Disorders
Keywords: mitoxantrone; neuromyelitis optica; relapse
MeSH Terms: conditions — Neuromyelitis Optica; Recurrence | interventions — Mitoxantrone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- MITO, annual relapse rate, safety (Other): For refractory NMO patients aged 18-55, the initial dose 12 mg/m2 mitoxantrone was administered over a five day course every 3 months for 2 years (a total of eight courses). The initial dose was reduced to 9 mg/m2 if the preinfusion white-blood-cell count was 3.0-3.99 ×109/L,and to 6 mg/m2 if the white-blood-cell count was 2.0-2.99 ×109/L. No infusion if the white-blood-cell count was less than 2.0×109/L. The initial dose was reduced to 10 mg/m2 for nonhaematological toxic effects of WHO grade 2-3. Subsequent dose after 3 month was reduced to 10 mg/m2 for infections that occurred within 3 weeks of a previous infusion accompanied by a white-blood-cell count below 2×109/L, or to 8 mg/m2 for infections accompanied by white-blood-cell count of less than 1×109/L.
  Interventions: Drug: Mitoxantrone

INTERVENTIONS:
Drug: Mitoxantrone — The treatment protocol consisted of 12 mg/m2 MITO intravenous infusions every 3 months for 2 years. Dosage was adjusted according to side effects.
  Other Names: Novantrone

SUMMARY:
The treatment protocol consisted of 12 mg/m2 MITO intravenous infusions every 3 months for 2 years. Dosage was adjusted according to side effects. Neurological assessment including the determination of the Expanded Disability Status Scale (EDSS) score and ophthalmologic evaluations were performed every 3 months and during relapses. Flow cytometric analysis, brain and spinal cord MRI was performed at baseline, 6, 12, 18, and 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Recurrent longitudinal myelitis (>3 segments of spinal cord involvement by MRI) with or without recurrent ON (unilateral or bilateral) but with normal brain MRI and positive serological NMO IgG antibody.
* Recurrent longitudinal myelitis (>3 segments of spinal cord involvement by MRI) with or without spatially limited brain lesion and positive serological NMO IgG antibody.
* NMO, fulfilled Wingerchuk 2006 Criteria for NMO.
* Patient presented at least 2 relapses during the 12 months preceding the start of mitoxantrone therapy, despite immunotherapies using corticosteroid, interferon beta, azathioprine, cyclophosphamide, Cyclosporin A, Mycophenolate Mofetil or a combination of these drugs
* Extended Disability Status Score 3-8.
* Normal range for white-blood-cell count (more than 4×109/L), neutrophil count (more than 2×109/L), and platelet count (more than 100×109/L).

Exclusion Criteria:

* Cardiac risk factors (e.g history of congestive heart failure and left ventricular ejection fraction (LVEF) < 50%
* Systemic diseases such as lupus, Sjogren's syndrome, anti-phospholipid antibody syndrome, sarcoidosis, rheumatoid arthritis, or vitamin B12 deficiency
* Previous treatment with mitoxantrone or anthracyclines
* Pregnant or planning to be pregnant
* Patients with severe liver disorders (WHO grade 4)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2009-03; Primary Completion 2014-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
annual relapse rate (ARR) | one year
  ARR is defined as the number of confirmed relapses in a year. The number of annual relapse rate was used as parameters of effectiveness and was compared between premitoxantrone and postmitoxantrone treatment during the follow-up period.
EDSS | six months
  Expanded Disability Status Scale (EDSS) scores was used as parameters of effectiveness and was compared between premitoxantrone and postmitoxantrone treatment during the follow-up period.

SECONDARY OUTCOMES:
Changes in LVEF | six months
  - Assessment of cardiac function: Changes in LVEF by transthoracic echocardiography and determination of cardiac side effects by ECG and by measurement of CK-MB, Troponin and BNP.
blood cell count | three months
  - Assessment of hematological system: Monitoring blood cell count regularly. Considering marrow puncture if necessary.
Flow cytometric analysis | six months
  Immunofluorescent staining of wholeblood samples were performed of blood drawing using antibodies against CD3/CD4/CD8/CD19/CD20/CD56 with isotype controls, followed by lysis of red blood cells and immediate acquisition and analysis by flow cytometry.

CONTACTS AND LOCATIONS:
Overall Officials: Huiqing Dong, Doctor, Principal Investigator — Department of Neurology, Xuanwu Hospital, Capital Medical University
Locations (1):
- Department of Neurology, Xuanwu Hospital, Capital Medical University, Beijing, Beijing Municipality, China

REFERENCES:
- [Background] Hartung HP, Gonsette R, Konig N, Kwiecinski H, Guseo A, Morrissey SP, Krapf H, Zwingers T; Mitoxantrone in Multiple Sclerosis Study Group (MIMS). Mitoxantrone in progressive multiple sclerosis: a placebo-controlled, double-blind, randomised, multicentre trial. Lancet. 2002 Dec 21-28;360(9350):2018-25. doi: 10.1016/S0140-6736(02)12023-X. PMID 12504397
- [Background] Neuhaus O, Kieseier BC, Hartung HP. Therapeutic role of mitoxantrone in multiple sclerosis. Pharmacol Ther. 2006 Jan;109(1-2):198-209. doi: 10.1016/j.pharmthera.2005.07.002. Epub 2005 Aug 10. PMID 16095713
- [Background] Kim SH, Kim W, Park MS, Sohn EH, Li XF, Kim HJ. Efficacy and safety of mitoxantrone in patients with highly relapsing neuromyelitis optica. Arch Neurol. 2011 Apr;68(4):473-9. doi: 10.1001/archneurol.2010.322. Epub 2010 Dec 13. PMID 21149806
- [Background] Weinstock-Guttman B, Ramanathan M, Lincoff N, Napoli SQ, Sharma J, Feichter J, Bakshi R. Study of mitoxantrone for the treatment of recurrent neuromyelitis optica (Devic disease). Arch Neurol. 2006 Jul;63(7):957-63. doi: 10.1001/archneur.63.7.957. PMID 16831964